CLINICAL TRIAL: NCT03532373
Title: Testing of a Tool to Elicit Patient Preferences for CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Duke University (Other); Brown University (Other); University of Texas at Austin (Other); Mayo Clinic (Other); Harvard University (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 46107; K23AR073307 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Carpal Tunnel; Carpal Tunnel Syndrome; Carpal Tunnel Syndrome Left; Carpal Tunnel Syndrome Right; Carpal Tunnel Syndrome Bilateral
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the intervention or control group
Masking Description: No masking will occur
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): None- normal care
- Intervention (Experimental): Patients will use a preference elicitation tool to determine their preferences for diagnosis and treatment of CTS
  Interventions: Other: Preference Elicitation tool

INTERVENTIONS:
Other: Preference Elicitation tool — A preference elicitation tool for carpal tunnel syndrome
  Arms: Intervention

SUMMARY:
This study will complete a randomized controlled trial to quantitatively measure patient decisional conflict (Decisional Conflict Scale) in 150 patients treated for CTS with the tool compared to 150 patients treated with standard care. The investigators hypothesize patients treated for CTS will have lower decisional conflict with the tool.

DETAILED DESCRIPTION:
The investigators will measure decisional conflict in 150 new patients being evaluated for CTS with the tool compared to 150 patients being evaluated for CTS with standard care. Those patients randomized to receiving the tool will use it to identify their preferences for certain attributes of care. Patients will then be presented with their preference data and the surgeon will have a discussion with the patient regarding CTS. Surgeons will have their standard discussion with the patients randomized to the standard care group (no tool). The tool will be operationalized on a Health Insurance Portability and Accountability Act compliant data platform, such as Qualtrics, and no identifiable data will be collected. De-identified data will be shared from study cites with our team at Stanford. This data will be backed up on a computer encrypted by Stanford.

ELIGIBILITY:
Inclusion Criteria:

* New patient
* English fluency and literacy
* Able to take informed consent
* clinical diagnosis of carpal tunnel syndrome

Exclusion Criteria:

* Prior diagnostic testing for carpal tunnel (nerve test, ultrasound)
* Prior carpal tunnel release
* Diagnosis of C5/6 radiculopathy (double crush)
* Peripheral neuropathy (ex: diabetic)
* Worker Compensation/EMG Required
* Symptoms of Cubital tunnel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Background] Zhang S, Vora M, Harris AH, Baker L, Curtin C, Kamal RN. Cost-Minimization Analysis of Open and Endoscopic Carpal Tunnel Release. J Bone Joint Surg Am. 2016 Dec 7;98(23):1970-1977. doi: 10.2106/JBJS.16.00121. PMID 27926678
- [Background] Atroshi I, Englund M, Turkiewicz A, Tagil M, Petersson IF. Incidence of physician-diagnosed carpal tunnel syndrome in the general population. Arch Intern Med. 2011 May 23;171(10):943-4. doi: 10.1001/archinternmed.2011.203. No abstract available. PMID 21606100
- [Background] Fajardo M, Kim SH, Szabo RM. Incidence of carpal tunnel release: trends and implications within the United States ambulatory care setting. J Hand Surg Am. 2012 Aug;37(8):1599-605. doi: 10.1016/j.jhsa.2012.04.035. Epub 2012 Jun 23. PMID 22727925
- [Background] Hageman MG, Kinaci A, Ju K, Guitton TG, Mudgal CS, Ring D; Science of Variation Group. Carpal tunnel syndrome: assessment of surgeon and patient preferences and priorities for decision-making. J Hand Surg Am. 2014 Sep;39(9):1799-1804.e1. doi: 10.1016/j.jhsa.2014.05.035. Epub 2014 Aug 1. PMID 25087865
- [Background] Oshima Lee E, Emanuel EJ. Shared decision making to improve care and reduce costs. N Engl J Med. 2013 Jan 3;368(1):6-8. doi: 10.1056/NEJMp1209500. No abstract available. PMID 23281971
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Alfandre D. Clinical Recommendations in Medical Practice: A Proposed Framework to Reduce Bias and Improve the Quality of Medical Decisions. J Clin Ethics. 2016 Spring;27(1):21-7. PMID 27045301
- [Background] Mulley AG, Trimble C, Elwyn G. Stop the silent misdiagnosis: patients' preferences matter. BMJ. 2012 Nov 8;345:e6572. doi: 10.1136/bmj.e6572. No abstract available. PMID 23137819
- [Background] Lang F, Floyd MR, Beine KL. Clues to patients' explanations and concerns about their illnesses. A call for active listening. Arch Fam Med. 2000 Mar;9(3):222-7. doi: 10.1001/archfami.9.3.222. PMID 10728107
- [Background] Johnson DC, Mueller DE, Deal AM, Dunn MW, Smith AB, Woods ME, Wallen EM, Pruthi RS, Nielsen ME. Integrating Patient Preference into Treatment Decisions for Men with Prostate Cancer at the Point of Care. J Urol. 2016 Dec;196(6):1640-1644. doi: 10.1016/j.juro.2016.06.082. Epub 2016 Jun 23. PMID 27346032
- [Background] Fraenkel L, Chodkowski D, Lim J, Garcia-Tsao G. Patients' preferences for treatment of hepatitis C. Med Decis Making. 2010 Jan-Feb;30(1):45-57. doi: 10.1177/0272989X09341588. Epub 2009 Jul 27. PMID 19636065
- [Background] Hageman MG, Bossen JK, Neuhaus V, Mudgal CS, Ring D; Science of Variation Group. Assessment of Decisional Conflict about the Treatment of carpal tunnel syndrome, Comparing Patients and Physicians. Arch Bone Jt Surg. 2016 Apr;4(2):150-5. PMID 27200394
- [Background] Kamal RN; Hand Surgery Quality Consortium. Quality and Value in an Evolving Health Care Landscape. J Hand Surg Am. 2016 Jul;41(7):794-9. doi: 10.1016/j.jhsa.2016.05.016. PMID 27374791
- [Background] Keith MW, Masear V, Amadio PC, Andary M, Barth RW, Graham B, Chung K, Maupin K, Watters WC 3rd, Haralson RH 3rd, Turkelson CM, Wies JL, McGowan R. Treatment of carpal tunnel syndrome. J Am Acad Orthop Surg. 2009 Jun;17(6):397-405. doi: 10.5435/00124635-200906000-00008. PMID 19474449
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240
- [Background] Graham B. The value added by electrodiagnostic testing in the diagnosis of carpal tunnel syndrome. J Bone Joint Surg Am. 2008 Dec;90(12):2587-93. doi: 10.2106/JBJS.G.01362. PMID 19047703
- [Background] Graham B. The diagnosis and treatment of carpal tunnel syndrome. BMJ. 2006 Jun 24;332(7556):1463-4. doi: 10.1136/bmj.332.7556.1463. No abstract available. PMID 16793786
- [Background] Graham B, Regehr G, Naglie G, Wright JG. Development and validation of diagnostic criteria for carpal tunnel syndrome. J Hand Surg Am. 2006 Jul-Aug;31(6):919-24. PMID 16886290
- [Background] Fowler JR, Cipolli W, Hanson T. A Comparison of Three Diagnostic Tests for Carpal Tunnel Syndrome Using Latent Class Analysis. J Bone Joint Surg Am. 2015 Dec 2;97(23):1958-61. doi: 10.2106/JBJS.O.00476. PMID 26631997
- [Background] Pulikkottil BJ, Schub M, Kadow TR, Wang W, Fowler JR. Correlating Median Nerve Cross-sectional Area With Nerve Conduction Studies. J Hand Surg Am. 2016 Oct;41(10):958-962. doi: 10.1016/j.jhsa.2016.08.018. PMID 27702467
- [Background] Flynn KE, Weinfurt KP, Seils DM, Lin L, Burnett CB, Schulman KA, Meropol NJ. Decisional conflict among patients who accept or decline participation in phase I oncology studies. J Empir Res Hum Res Ethics. 2008 Sep;3(3):69-77. doi: 10.1525/jer.2008.3.3.69. PMID 19122780
- [Background] Hyman DJ, Pavlik VN, Greisinger AJ, Chan W, Bayona J, Mansyur C, Simms V, Pool J. Effect of a physician uncertainty reduction intervention on blood pressure in uncontrolled hypertensives--a cluster randomized trial. J Gen Intern Med. 2012 Apr;27(4):413-9. doi: 10.1007/s11606-011-1888-1. Epub 2011 Oct 27. PMID 22033742
- [Background] Wittink MN, Cary M, Tenhave T, Baron J, Gallo JJ. TOWARDS PATIENT-CENTERED CARE FOR DEPRESSION: CONJOINT METHODS TO TAILOR TREATMENT BASED ON PREFERENCES. Patient. 2010;3(3):145-157. doi: 10.2165/11530660. PMID 20671803
- [Background] Baker LC, Bundorf MK, Kessler DP. Patients' preferences explain a small but significant share of regional variation in medicare spending. Health Aff (Millwood). 2014 Jun;33(6):957-63. doi: 10.1377/hlthaff.2013.1184. PMID 24889944
- [Background] Hampson LA, Allen IE, Gaither TW, Lin T, Ting J, Osterberg EC, Wilson L, Breyer BN. Patient-centered Treatment Decisions for Urethral Stricture: Conjoint Analysis Improves Surgical Decision-making. Urology. 2017 Jan;99:246-253. doi: 10.1016/j.urology.2016.07.053. Epub 2016 Sep 16. PMID 27645527

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients use a preference elicitation tool to determine their preferences for diagnosis and treatment of CTS
Period: Overall Study
Arm/Group | Control | Intervention
Started | 19 | 30
Completed | 19 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 19 | 30 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (17.9) | 54.6 (18.5) | 55.5 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 12 | 18 | 30
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 30 | 49
CTS-6 [Mean (Standard Deviation); unit: units on a scale] — Score range: 0 to 26 (higher scores indicate more severe carpal tunnel symptoms)
  units on a scale | 18.2 (5.9) | 18.1 (3.8) | 18.2 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale
Description: The Decisional Conflict Scale measures uncertainty in choosing options; modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. The survey consists of 16 statements with 5 response categories. Scoring: total scale-0 (no decisional conflict) to 100 (extreme decisional conflict). Lower values indicate lower decisional conflict- i.e. a better outcome for use of the tool. Calculation: Summed, divided by # of items, multiplied by 25
Time Frame: Immediately after using tool (up to 5 minutes to complete survey)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 30
score on a scale | 1.77 (4.6) | 4.41 (10.3)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/30
Other Adverse Events (participants affected / at risk) | 0/19 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03532373/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03532373/ICF_001.pdf